CLINICAL TRIAL: NCT03770065
Title: A Phase II, Open-label, Single-Centre, Randomized, Cross-over, Exploratory Study on Two Different Doses of VML-0001, the Base Formulation of Viramal's pH Regulating and Vaginal Moisturizing Cream, on the Effects on Vaginal pH in Healthy Post-Menopausal Women
Brief Title: Exploratory Study on Two Different Doses of VML-0001 on the Effects on Vaginal pH in Healthy Post-Menopausal Women
Status: Completed | Type: Observational
Sponsor: Viramal Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: VML-0001-003
Record Dates: First submitted 2018-12-04; First posted 2018-12-10 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Vaginal Atrophy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A
  Interventions: Device: VML-0001
- Group B
  Interventions: Device: VML-0001

INTERVENTIONS:
Device: VML-0001 — Medical device

SUMMARY:
The study is designed to determine the effect on vaginal pH and the duration of action measured on the ability of the base formulation to reduce the vaginal pH

ELIGIBILITY:
Inclusion Criteria:

* be greater than 45 years
* no positive findings on screening gynaecological examination
* negative smear test within the last 5 years

Exclusion Criteria:

* has signs of vaginal infection
* has evidence of alcohol abuse
* has used hormonal replacement therapy in three months prior to study entry

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Healthy post-menopausal women
Study Population: Healthy Post-Menopausal women
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-04-08 (Actual)

PRIMARY OUTCOMES:
To determine the duration of action measured on the ability of VML-0001 (base formulation) to reduce vaginal pH. | 7-14 days
  The Vaginal pH will be measured daily for 7 days after single dose of VML-0001 using pH kits.

CONTACTS AND LOCATIONS:
Overall Officials: James Murray, MD, Principal Investigator — Doctor
Locations (1):
- Medical Affiliated Research Center, Inc. (MARC), Huntsville, Alabama, United States